CLINICAL TRIAL: NCT01286714
Title: Assessment of Fistula Closure by OTSC Clip After Bariatric Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique Hopitaux De Marseille (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2010-A01210-39; 2010-21 (Other: AP HM)
Record Dates: First submitted 2011-01-28; First posted 2011-01-31 (Estimated); Last update posted 2014-08-29 (Estimated); Status verified 2014-08

CONDITIONS: Bariatric Surgery (Sleeve Gastrectomy )

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- clips OST (Experimental)
  Interventions: Device: CLIP OST

INTERVENTIONS:
Device: CLIP OST

SUMMARY:
Anastomotic fistula following bariatric surgery are lifethreatening complication with a 37.5% mortality rate. All the modalities for bariatric surgery are involved in this type of complication, but Sleeve gastrectomy is the main surgery responsible for the frequency and the severity of the fistula. The management of this complication is still controversial and potentially lethal. The average number of endoscopic sessions was 4 (range 2-11). The closure could be obtained within a mean time of 88 days (range 6-216 days). Therefore endoscopic management has to be improved to reduce the duration of the treatment and the number of endoscopic sessions. OTSC clips could help to improve the endoscopic management because of a more prehensive, deeper and larger suture area.

ELIGIBILITY:
Inclusion Criteria:

* age upper to 18 years
* surgery bariatrique typical Sleeve
* presence of one or two fistulas < 1 cm, beforehand drained and without sepsis evolutionary
* signature of the consent

Exclusion Criteria:

* surgery bariatrique other one than Sleeve
* refusal of the patient of this endoscopic repeated coverage(care) requiring several sessions of endoscopies under AG with hospitalizations
* Current Sepsis
* not drained cavity
* Absence of signed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2011-01; Primary Completion 2013-09 (Actual); Study Completion 2013-09 (Actual)

PRIMARY OUTCOMES:
The efficacity of closure of fistulas by clips ovesco | 12 months

SECONDARY OUTCOMES:
The efficacity of the suture in 3 months of these complex refractory fistulas | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: BERNARD BELAIGUES, Study Director — Assistance Publique hôpitaux de Marseille
Locations (1):
- Assistance Publique Hopitaux de Marseille, Marseille, France